CLINICAL TRIAL: NCT05159479
Title: Defining Robust Predictors of Chemotherapy Related Cardiotoxicity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 140342
Record Dates: First submitted 2021-12-01; First posted 2021-12-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cardiotoxicity; Gastrointestinal Neoplasms
Keywords: Fluoropyrimidine; Cardiotoxicity; Cardio-oncology
MeSH Terms: conditions — Cardiotoxicity; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational prospective cohort study designed for patients with gastrointestinal cancers receiving a fluoropyrimidine based chemotherapy regimen.

DETAILED DESCRIPTION:
All enrolled participants will undergo baseline cardiovascular risk assessment (using QRISK3 and SCORE 2 risk calculators), cardiac, oncological and medication history. All participants will have serial cardiac symptom assessment, 12 lead ECG and cardiac biomarker assessments(high sensitivity troponin T and NT pro BNP) at baseline, on completion of the first cycle of treatment and post completion of treatment. Participants will be followed up for the development of cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Consented to receive fluoropyrimidine chemotherapy for GI malignancies (gastro-oesophageal, colorectal, pancreatic)
* Capacity to provide consent

Exclusion Criteria:

* Age <18
* Lacking capacity to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from secondary or tertiary care centres from oncology clinics. Participants included will be undergoing chemotherapy in the neoadjuvant, adjuvant and palliative setting.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of fluoropyrimidine induced cardiotoxicity (FIC) | 12 months
  Fluoropyrimidine induced cardiotoxicity defined as a composite of:
  * Types 1-3 myocardial infarction with troponin >99th percentile upper limit,
  * Incident myocardial ischaemia (chest pain with or without new inducible perfusion abnormality on perfusion cardiac MRI,
  * Myocarditis (diagnosed as per European Society of Cardiology Consensus statement)
  * Incident heart failure (HF) diagnosis (symptoms with raised N-terminal pro-B-type natriuretic peptide (NTproBNP )> 400pg/ml or HF hospitalisation),
  * Incident arrhythmia (excluding isolated ectopy) or sudden cardiac death.
Relationship of baseline cardiovascular risk with FIC | 12 months
  Baseline cardiovascular risk assessed using QRISK3 cardiovascular risk calculator
Relationship of baseline cardiovascular risk with FIC | 12 months
  Baseline cardiovascular risk assessed using SCORE2 cardiovascular risk calculator

SECONDARY OUTCOMES:
Change in cardiac biomarkers (high sensitivity troponin T) | Assessed at baseline pre chemotherapy, after cycle 1 chemotherapy (46 hours for patients on 5-FU and day 14 for patients on capecitabine) and at end of treatment (at 6 weeks post completion)
Change in cardiac biomarkers (NT pro BNP) | Assessed at baseline pre chemotherapy, after cycle 1 chemotherapy (46 hours for patients on 5-FU and day 14 for patients on capecitabine) and at end of treatment (at 6 weeks post completion)
Cardiovascular symptom assessment | Assessed at baseline pre chemotherapy, after cycle 1 chemotherapy (46 hours for patients on 5-FU and day 14 for patients on capecitabine) and at end of treatment (at 6 weeks post completion)
  Using modified seattle angina questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomews Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No